CLINICAL TRIAL: NCT06864416
Title: Comparative Study Between Dexmedetomidine and Fentanyl as Adjuvants to Bupivacaine in Femero Sciatic Block for Below Knee Surgery
Brief Title: Comparative Study Between Dexmedetomidine and Fentanyl as Adjuvants to Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS199/2024
Record Dates: First submitted 2025-02-14; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (dexmedetomidine group ) (Active Comparator): the sciatic and femoral nerve blocks will be achieved using A 40 ml mixture consisting of 0.25% bupivacaine and 1 µ/kg dexmedetomidine.
  Interventions: Drug: dexmedetomidine as adjuvant to bupivacaine
- group (fentanyl group ) (Active Comparator): the sciatic and femoral nerve blocks will be achieved using A 40 ml mixture consisting of 0.25% bupivacaine with 1 µg/kg of fentanyl.
  Interventions: Drug: Fentanyl as adjuvant to bupivacaine

INTERVENTIONS:
Drug: dexmedetomidine as adjuvant to bupivacaine — the efficacy of addition of dexmedetomidine as adjuvants to bupivacaine in femorosciatic nerve block
  Other Names: adjuvants to local anesthetics
  Arms: group (dexmedetomidine group )
Drug: Fentanyl as adjuvant to bupivacaine — the efficacy of addition of fentanyl as adjuvants to bupivacaine in femorosciatic nerve block
  Other Names: adjuvants to local anesthetics
  Arms: group (fentanyl group )

SUMMARY:
Combined femoral and sciatic nerve block provides surgical anesthesia with better cardiorespiratory stability as compared to the spinal anesthesia blockade which has side effects of hypotension, bradycardia, meningitis, post dural puncture headache, hematoma, and neurological deficit

DETAILED DESCRIPTION:
Combined femoral and sciatic nerve block provides surgical anesthesia with better cardiorespiratory stability as compared to the spinal anesthesia blockade which has side effects of hypotension, bradycardia, meningitis, post dural puncture headache, hematoma, and neurological deficit, Adjuvants are those drugs which, when co-administered with local anesthetic agents, may improve the speed of onset and duration of analgesia and counteract disadvantageous effects of local anesthetics. By adding these adjuvants, the dose of local anesthetics like bupivacaine can be reduced, thereby reducing its side effects like myocardial depression, hypotension, bradycardia, heart block, and ventricular arrhythmias. Based on "Combination Wisdom", the use of adjuvants to local anesthetics has been promoted a lot .A wide variety of drugs have been used for both neuraxial and peripheral nerve blocks, and the most commonly used drug as adjuvant is the fentanyl .

The addition of dexmedetomidine during US-guided combined femoral and sciatic block for below knee surgery was associated with a prolonged duration of analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years.
* American Society of Anesthesiologists (ASA) physical status I-II,
* Scheduled for elective surgery below the knee.

Exclusion Criteria:

* Allergies to used medications.
* Coagulopathy.
* Septic patients.
* Neurological disease.
* Respiratory or cardiac disease.
* Diabetes mellitus.
* Patients' refusal to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue score assessment | 6 hours from performing the block
  Score range from zero to ten , lower score indicate accepted out come

SECONDARY OUTCOMES:
The time of first analgesics required | Immediately after the end of the surgery and for 48 hours
  analgesics requirements

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, abbasia, Cairo, Egypt